CLINICAL TRIAL: NCT01213771
Title: Health and Coping Prior to Ovarian Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other); Aarhus University Hospital (Other); Danish Cancer Society (Other)
Responsible Party: Lene Seibæk, Aarhus Univerity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LS2008
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Health and Coping Undergoing Ovarian Cancer Surgery.; Cancer Rehabilitation
Keywords: Preoperative; Intervention; Support; Care
MeSH Terms: interventions — Preoperative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative care 2009 (No Intervention): Patients are receiving the usual care
  Interventions: Procedure: Preoperative preparation 2010

INTERVENTIONS:
Procedure: Preoperative preparation 2010 — Preoperative optimisation Supportive care LEAN in patient pathways
  Other Names: Preoperative care

SUMMARY:
Background Denmark has a record-high incidence of, and mortality rate for, ovarian cancer. There are 600 new cases of ovarian cancer each year. In 2008 the state issued a guarantee of early diagnosis and treatment of all cases of suspected cancer, and surgical treatment has been centralised and standardised in fast track programmes. However, the investigators do not know how women with ovarian cancer experience the period prior to surgery and how they can optimally prepare for treatment and care.

Aim The two principal aims of the study are to describe health and coping in Danish women surgically treated for ovarian cancer; and to examine to what extent it is possible, from both a patient and professional perspective, to improve the health and everyday life of patients with ovarian cancer.

Materials and methods The study is conducted within the scientific theoretical framework of hermeneutics, involving the overall concepts of health promotion and rehabilitation. The study will be carried out in 4 stages between September 2008 and September 2011. Stage 1: A health-related characterisation of Danish women with ovarian cancer through a registration process. Stage 2: Qualitative research interviews with patients, to gain knowledge about spontaneous preoperative coping strategies and resources.

Stage 3: The preoperative preparation programme will be developed and clinically tested. The effect of participation will be measured by self-assessed health and coping before and after surgery. The study period runs from the time the decision is taken to operate until eight weeks after discharge. The study takes place at the Department of Gynaecology at Aarhus University Hospital, Skejby in Denmark, which is a regional centre of surgical treatment of gynaecological cancer.

Results The study provides insight into the preoperative coping strategies and general health of Danish women suffering from ovarian cancer. The development and testing of the preoperative preparation programme contributes to knowledge about optimisation of preoperative preparation. This might have a positive impact on the participants' general health and level of functioning during their treatment. Furthermore, the project contributes to knowledge of the preoperative coping strategies and experiences of (female) cancer patients in general.

DETAILED DESCRIPTION:
Supervisors Lise Hounsgaard, Associate Professor, PhD, Research Unit of Nursing, Institute of Clinical Research, Faculty of Health Sciences, University of Southern Denmark. Lone Kjeld Petersen, Consultant, DMSc. and Jan Blaakær, Consultant, DMSc.Department of Gynaecology and Obstetrics Y, Aarhus University Hospital, Skejby.

Funding Faculty of Health Sciences, University of Southern Denmark. Department of Gynaecology and Obstetrics Y, Aarhus University Hospital, Skejby. The Research Foundation of Health Science in Central Denmark Region. The Research Foundation of Aarhus University Hospital, Skejby. The Hede Nielsen Foundation. The Danish Cancer Society, Psychosocial Research Committee. Tha Danish Nurses organisation

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing surgery on the suspicion of an ovarian malignancy

Exclusion Criteria:

* Mental disease, not being able to understand Danish,

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
SF 36 | The day before surgery and 8 weeks after surgery
  The peri-operative period

CONTACTS AND LOCATIONS:
Overall Officials: Lise Hounsgaard, ass. prof., Study Chair — University of Southern Denmark
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark